CLINICAL TRIAL: NCT01348191
Title: Detection of Thyrotrophin Receptor in Human Myometrium
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Stichting PAMM (Unknown); Tilburg University (Other); Erasmus Medical Center (Other); Eindhoven University of Technology (Other)
Responsible Party: Principal Investigator, S.Kuppens, MD, Phd, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL36261.060.11
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Thyrothrophin Receptor in Myometrium Tissue
Keywords: Thyrotrophin; Pregnancy; Human myometrium; Relaxation; Contractility
MeSH Terms: interventions — Thyrotropin; Myocardial Contraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy of human myometrium
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elective caesarean section: Population: ten pregnant women, scheduled for elective caesarean section with a term pregnancy ( > 37 weeks).
  Inclusion criteria
  * Elective caesarean section
  * Term pregnancy > 37 weeks
  * Age > 18 years
  Exclusion criteria
  * Previous caesarean scar
  * Gestational age < 37 weeks
  * Maternal temperature > 37.8 degrees Celsius
  * Meconium stained liquor
  * Foetal distress
  * Maternal diabetes
  * Seropositivity
  * Use of thyroid medication
  * Maternal thyroid disease
  * Age < 18 years
  Interventions: Procedure: Myometrial biopsy

INTERVENTIONS:
Procedure: Myometrial biopsy — At caesarean section, after birth of the baby but before closure of the uterus, a biopsy from the upper lip of the incision in the lower uterine segment will be taken. This biopsy will measure approximately 2x50mm.
  Other Names: Thyrotrophin; Myometrium; Relaxation; Contractility; Conductance; Electropotentials

SUMMARY:
It has been recognized for many decades that high thyrotrophin (TSH) levels in pregnant women are associated with poor obstetric outcome. Also, there is evidence that high TSH is related to fetal position at term, including breech which in turn is associated with obstetric complications.

However, the mechanism behind remains to be elucidated.

The current project is of basic-fundamental nature. It is used to better understand basis physiological processes. As in many other studies of similar basic nature, few numbers are always included.

If a TSH receptor will be detected, future randomized controlled trials (RCT) might be worthwhile with large numbers of women who will be treated with thyroxine to possibly prevent abnormal fetal position during normal pregnancy.

The aim of the current study is to evaluate whether a TSH receptor can be demonstrated in human myometrium. If so, the pathophysiology of high TSH in relation to obstetric outcome will become more clear. Furthermore, the aim is to test the myometrium in vitro for its relaxation and contractility and for the conductance of electropotentials.

DETAILED DESCRIPTION:
It has been recognized for many decades that high thyrotrophin (TSH) levels in pregnant women are associated with poor obstetric outcome. Also, there is evidence that high TSH is related to fetal position at term, including breech which in turn is associated with obstetric complications.

However, the mechanism behind remains to be elucidated. It has been shown that high TSH affects relaxation and contraction of the smooth muscle in large blood vessels in human. In animals, there is some evidence that TSH interferes with uterine contractility. Although a TSH receptor has been demonstrated outside the thyroid in bone, brain and heart, so far no research on a possible TSH receptor in human uterine tissue has been published.

The current study is a pilot study in which in a limited number of participants (pregnant women, n=10) during elective Caesarean section a uterine specimen will be collected for analysis in a immune-laboratory.

Another part of the specimen will be analysed in a technical laboratory(Technical University of Eindhoven)for analysing the relaxation and contractility of the myometrium and for studying the conductance of electropotentials.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean section
* Term pregnancy > 37 weeks
* Age > 18 years

Exclusion Criteria:

* Previous caesarean scar
* Gestational age < 37 weeks
* Maternal temperature > 37.8 degrees Celsius
* Meconium stained liquor
* Foetal distress
* Maternal diabetes
* Seropositivity
* Use of thyroid medication
* Maternal thyroid disease
* Age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women (n=10) with a term ( > 37 weeks) baby, who are scheduled for elective caesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Thyrothrophin receptor | three months
  Immunodetection of Thyrothrophin receptor in myometrium tissue

SECONDARY OUTCOMES:
electropotentials in myometrium and relaxation and contractility | Three months
  Investigation of relaxation and contractility of myometrium. Conductance of electropotentials of myometrium tissue

CONTACTS AND LOCATIONS:
Overall Officials: simone M Kuppens, MD,PhD, Principal Investigator — Catharina-ziekenhuis, Eindhoven, the Netherlands; Victor J Pop, MD,PhD,Prof, Study Director — University of Tilburg, Department of Medical and Neuropsychology
Locations (4):
- Netherlands (4):
  - Catharina-hospital, Eindhoven, North Brabant
  - Eindhoven University of Technology, Eindhoven, North Brabant
  - University of Tilburg, Tilburg, North Brabant
  - Erasmus MC, Rotterdam, South Holland

REFERENCES:
- [Background] Potter SM, Astbury K, Morrison JJ. Effects of thyrotropin-releasing hormone on human myometrium and umbilical vasculature in vitro. Am J Obstet Gynecol. 2004 Jan;190(1):246-51. doi: 10.1016/s0002-9378(03)00853-6. PMID 14749667
- [Background] Oner J, Oner H. Immunodetection of thyroid hormone receptor (alpha1/alpha2) in the rat uterus and oviduct. Acta Histochem Cytochem. 2007 Jul 3;40(3):77-81. doi: 10.1267/ahc.06026. PMID 17653299
- [Background] Heemstra KA, van der Deure WM, Peeters RP, Hamdy NA, Stokkel MP, Corssmit EP, Romijn JA, Visser TJ, Smit JW. Thyroid hormone independent associations between serum TSH levels and indicators of bone turnover in cured patients with differentiated thyroid carcinoma. Eur J Endocrinol. 2008 Jul;159(1):69-76. doi: 10.1530/EJE-08-0038. Epub 2008 Apr 7. PMID 18390987
- [Background] Peeters RP, van der Deure WM, Visser TJ. Genetic variation in thyroid hormone pathway genes; polymorphisms in the TSH receptor and the iodothyronine deiodinases. Eur J Endocrinol. 2006 Nov;155(5):655-62. doi: 10.1530/eje.1.02279. PMID 17062880
- [Background] Kuppens SM, Kooistra L, Wijnen HA, Crawford S, Vader HL, Hasaart TH, Oei SG, Pop VJ. Maternal thyroid function during gestation is related to breech presentation at term. Clin Endocrinol (Oxf). 2010 Jun;72(6):820-4. doi: 10.1111/j.1365-2265.2009.03729.x. Epub 2009 Oct 15. PMID 19832853
- [Background] Kooistra L, Kuppens SM, Hasaart TH, Vader HL, Wijnen HA, Oei SG, Pop VJ. High thyrotrophin levels at end term increase the risk of breech presentation. Clin Endocrinol (Oxf). 2010 Nov;73(5):661-5. doi: 10.1111/j.1365-2265.2010.03846.x. PMID 20718770